CLINICAL TRIAL: NCT03822364
Title: A Randomized Study of the Safety, Tolerability, and Pharmacokinetics of AZ-009 (Staccato Apomorphine) in Healthy Volunteers and the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZ-009 in Subjects With Parkinson's Disease
Brief Title: Staccato Apomorphine Single and Multi Dose PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-009-101
Record Dates: First submitted 2018-12-18; First posted 2019-01-30 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2018-12

CONDITIONS: Parkinson Disease
Keywords: apomorphine; aerosol
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A 3 part study including: A) Single Dose Crossover in Healthy Volunteers, B) Single Ascending Dose with placebo control in Healthy Volunteers, and C) Single Ascending Dose with placebo control in Subjects with Established Parkinson's Disease
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (14):
- A-1 (009-1 -> active comparator) (Experimental): Part A, Arm 1 (Inhaled apomorphine, Dose 1 followed by commercially available active comparator)
  Interventions: Drug: 009-1; Drug: active comparator
- A-2 (active comparator -> 009-1) (Experimental): Part A, Arm 2 (commercially available active comparator followed by Inhaled apomorphine, Dose 1)
  Interventions: Drug: 009-1; Drug: active comparator
- B-1a (009-2) (Experimental): Part B, Arm 1 (Inhaled apomorphine, Dose 2)
  Interventions: Drug: 009-2
- B-1p (009-0) (Placebo Comparator): Part B, Arm 1 (Inhaled placebo)
  Interventions: Drug: 009-0
- B-2a (009-3) (Active Comparator): Part B, Arm 2 (Inhaled apomorphine, Dose 3)
  Interventions: Drug: 009-3
- B-2p (009-0) (Placebo Comparator): Part B, Arm 2 (Inhaled placebo)
  Interventions: Drug: 009-0
- B-3a (009-4) (Experimental): Part B, Arm 3 (Inhaled apomorphine, Dose 4)
  Interventions: Drug: 009-4
- B-3p (009-0) (Placebo Comparator): Part B, Arm 3 (Inhaled placebo)
  Interventions: Drug: 009-0
- C-1a (009-3) (Experimental): Part C, Arm 1 (Inhaled apomorphine, Dose 3)
  Interventions: Drug: 009-3
- C-1p (009-0) (Placebo Comparator): Part C, Arm 1 (Inhaled placebo)
  Interventions: Drug: 009-0
- C-2a (009-4) (Experimental): Part C, Arm 2 (Inhaled apomorphine, Dose 4)
  Interventions: Drug: 009-4
- C-2p (009-0) (Placebo Comparator): Part C, Arm 2 (Inhaled placebo)
  Interventions: Drug: 009-0
- C-3a (009-5) (Experimental): Part C, Arm 3 (Inhaled apomorphine, Dose 5)
  Interventions: Drug: 009-5
- C-3p (009-0) (Placebo Comparator): Part C, Arm 3 (Inhaled placebo)
  Interventions: Drug: 009-0

INTERVENTIONS:
Drug: 009-1 — Inhaled apomorphine via Staccato aerosol, Dose 1
  Arms: A-1 (009-1 -> active comparator); A-2 (active comparator -> 009-1)
Drug: active comparator — commercially available apomorphine injector
  Arms: A-1 (009-1 -> active comparator); A-2 (active comparator -> 009-1)
Drug: 009-0 — Inhaled placebo via Staccato device
  Arms: B-1p (009-0); B-2p (009-0); B-3p (009-0); C-1p (009-0); C-2p (009-0); C-3p (009-0)
Drug: 009-2 — Inhaled apomorphine via Staccato aerosol, Dose 2
  Arms: B-1a (009-2)
Drug: 009-3 — Inhaled apomorphine via Staccato aerosol, Dose 3
  Arms: B-2a (009-3); C-1a (009-3)
Drug: 009-4 — Inhaled apomorphine via Staccato aerosol, Dose 4
  Arms: B-3a (009-4); C-2a (009-4)
Drug: 009-5 — Inhaled apomorphine via Staccato aerosol, Dose 5
  Arms: C-3a (009-5)

SUMMARY:
This study will be conducted in 3 parts. A) compare the pharmacokinetics (PK) of a single dose of AZ-009 with that of a therapeutically-relevant dose of a commercially available apomorphine injector in healthy volunteers; B) ascending doses of active drug in healthy volunteers; and C) examine the tolerability, safety, and PK of AZ-009 in subjects with established Parkinson's disease.

DETAILED DESCRIPTION:
This study will be conducted in 3 parts. Parts A and B will be conducted in healthy volunteers and Part C will be conducted in subjects with established Parkinson's disease. The primary objectives for each part are as follows.

Part A: To compare the pharmacokinetics of a single low dose of AZ-009 with that of a therapeutically-relevant dose a commercially available apomorphine injector in healthy volunteers.

Part B: To examine the tolerability and safety of AZ-009 of single ascending doses of active drug in healthy volunteers while; and to characterize the pharmacokinetics of single ascending doses of AZ-009 in healthy volunteers

Part C: To examine the tolerability, safety, and pharmacokinetics of AZ-009 in subjects with established Parkinson's disease and to identify optimal doses to bring into multiple ascending dose safety and efficacy studies; and to assess the usability of AZ-009 in subjects with Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females between 18 and 60 years of age, inclusive at the time of signing the informed consent document.
* Body weight ≥ 50 kg and BMI within the range of 18 to 32 kg/m2.
* Willing and able to be confined at the clinical research center for the study period and adhere to overall study visit schedule, procedures and other protocol requirements.
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.

Exclusion Criteria:

* Any significant medical condition, psychiatric illness or history of depression that could, in the investigator's opinion, compromise the subject's safety or interfere with the completion of this protocol.
* History of clinically significant central nervous system, cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal conditions including gastric bypass or other weight loss surgical procedure; or history of such conditions that, in the opinion of the investigator, may place the subject at an unacceptable risk as a participant in this trial.
* Use of non-prescription medications within 5 days prior to the first dose of study drug.
* Use of medication that is inhibitor or inducer of CYP450-3A4/5 within 3 days of dosing.
* Consumption of grapefruit, grapefruit juice, star fruit, oranges, orange juice, Seville oranges, within 3 days prior to administration of study drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
A-Relative bioavailability of inhaled Staccato apomorphine dose compared to the subcutaneous administration | 24 hours
  Relative bioavailability of inhaled Staccato apomorphine compared to active comparator injection based on the Geometric Least Squares Mean Ratio of AUCinf for all subjects completing the crossover part of the trial
B-Dose Proportionality by Power Analysis of AUCinf | 24 hours
  Dose proportionality of inhaled Staccato apomorphine AUCinf across all doses administered in the single ascending dose portions of the study (Parts B and C) using a power model [regression of log(AUCinf) versus log(dose)]

CONTACTS AND LOCATIONS:
Overall Officials: Geert J Groeneveld, MD, PhD, Principal Investigator — Center for Human Drug Research (The Netherlands)
Locations (1):
- Center for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided